CLINICAL TRIAL: NCT07252999
Title: Transection Versus Reduction of Hernia Sac in Open Pediatric Inguinal Hernia Repair: A Randomized Controlled Trial Study
Brief Title: Comparison of Outcomes of Hernia Sac Transection and Sac Reduction in Open Pediatric Inguinal Hernia Repair in Ramathibodi Hospital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Piyanuch Lormuangthong (Other)
Collaborators: Ramathibodi Hospital (Other)
Responsible Party: Sponsor-Investigator, Piyanuch Lormuangthong, Principle investigator, Mahidol University
Organization: Mahidol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURA2025/684
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Inguinal Hernia Repair
Keywords: hernia sac transection; hernia sac reduction; open inguinal hernia repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hernia sac transection (Experimental): Patients who underwent open inguinal hernia surgery using hernia sac transection technique.
  Interventions: Procedure: Hernia sac transection
- Hernia sac reduction (Active Comparator): Patients who underwent open inguinal hernia surgery using hernia sac reduction technique.
  Interventions: Procedure: hernia sac reduction

INTERVENTIONS:
Procedure: Hernia sac transection — After administering anesthesia, a standard open inguinal hernia surgery typically was performed by the surgeon. Open inguinal hernia surgery using hernia sac transection technique. Other practices for the patient were as per standard care, including examination, diagnosis, treatment and follow-up.
  Arms: Hernia sac transection
Procedure: hernia sac reduction — After administering anesthesia, a standard open inguinal hernia surgery typically was performed by the surgeon. Open inguinal hernia surgery using hernia sac reduction technique. Other practices for the patient were as per standard care, including examination, diagnosis, treatment and follow-up.
  Arms: Hernia sac reduction

SUMMARY:
The goal of this clinical trial is to learn if hernia sac transection works to treat pediatric inguinal hernia. Researchers will compare hernia sac transection to hernia sac reduction (traditional inguinal hernia repair) to see outcome in 6 months. Visit the clinic at week1, month3, month 6 for follow-up.

DETAILED DESCRIPTION:
An inguinal hernia is a common condition in children where abdominal contents push through a weak spot in the abdominal wall into the groin area. Normally, when the testicles move from the abdomen into the scrotum, the peritoneal lining is pulled downward with them through the inguinal canal. The testicles are fully descended into the scrotum at about eighth months of gestation. Afterward, the opening created by this pouch closes and dissolves. The persistence of this inguinal canal, which should have closed spontaneously, is a common cause of hernias in children, with an incidence of 3.5-5% and it increases up to 44-55% in premature infants. Inguinal hernias often require surgical repair due to the risk of complications like bowel obstruction, which occurs in a significant percentage of cases with an incidence of 3-16%. Open surgery remains the most common method for inguinal hernias. A study by Chukwubuike KE et al. found that pediatric inguinal hernia repair had a postoperative complication rate of 9.9%. The most common complications were scrotal edema, scrotal hematoma, wound infection, hernia recurrence, testicular atrophy และsensory disturbance in the groin region.

Laparoscopic hernia surgery has become more widely used since the first operation in 1993. In this procedure, the hernia sac is cut open and the patent processus vaginalis is used to tighten the internal inguinal ring to prevent future hernias. The purse-string technique is used to close the opening of the internal ring without removing the hernia sac. Laparoscopic surgery offers faster recovery and less risk of spermatic cord injury, with similar operative times and shorter hospital stays compared to open surgery. However, it requires a higher initial cost and the expertise of a surgeon experienced in the procedure.

In a study by Kelly Dreuning, Laparoscopic versus open pediatric inguinal hernia repair: state of the art comparison and future perspectives from a meta-analysis, laparoscopic and open hernia repairs were performed in 375 and 358 patients, respectively. There was no difference in recurrence between the two groups.

Open hernia repair is still used for pediatric patients at Ramathibodi Hospital in order to remove the hernia sac from the spermatic cord. It is a complicated procedure, especially when dealing with big hernias. In a study by Roberto Cirocchi et al., Comparison of hernia sac transection and full sac reduction for the treatment of inguinal hernia: A systematic review and meta-analysis of clinical trials, 1,824 patients were included in the systematic review and meta-analysis of clinical trials which comprised 12 randomized controlled trials (RCTs) and 3 controlled clinical trials (CCTs). Nine hundred and thirty-five of these 1,824 patients had hernia sac transection, and nine hundred and sixty-six had hernia sac reduction. The study found that the two techniques were similar in terms of primary and secondary outcomes, even though hernia sac reduction might lead to a lower, albeit not statistically significant, recurrence rate.

The study by Mohamed Ali Chaouch et al., A systematic review and meta-analysis of hernia sac management in laparoscopic groin hernia mesh repair: reduction or transection, is a systematic review and meta-analysis (PRISMA) study which included 6 studies with a total of 2,941 patients: 821 in the transection group and 2,120 in the reduction group. It was found that the transection group had a significantly lower rate of postoperative seroma than the reduction group (OR = 1.71; 95% CI [1.22, 2.39], p = 0.002). However, there was no significant difference between the two groups in operative time (MD = -4.39; 95%CI [-13.62, 4.84], p = 0.35) and recurrence rate (OR = 2.70; 95%CI [0.50,14.50], p = 0.25)

The aforementioned information indicates that research has been done on the rates of complications following hernia surgery involving the excision of the hernia sac by reduction and transection. However, as of now, there are no conclusive findings about laparoscopic surgery. Thus, this study aimed to assess the rates of complications in pediatric patients who underwent open hernia surgery using reduction and transection techniques.

ELIGIBILITY:
Inclusion Criteria:

* Male pediatric patients under 18 years old
* Patients who underwent open inguinal hernia surgery on the affected side by a pediatric surgeon
* Patients who had follow-up after inguinal hernia surgery at Ramathibodi Hospital or phone follow-up (Telemed) for 6 months
* Patients who agree to participate in the study by signing an informed consent form

Exclusion Criteria:

* Preterm infants
* Inguinal hernia patients with strangulated hernia
* Patients with non-communicating hydrocele
* Patients who had follow-up at another hospital after inguinal hernia surgery
* Patients who refused to participate in the study or withdrawn

Ages: 1 Day to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reactive hydrocele | post-operative follow-up at week1, month3, month6
  Number of Participants with diagnosed through a physical examination that includes a transillumination test, where a soft, fluid-filled mass in the scrotum will glow with a soft, transparent light
Scrotal hematoma | post-operative follow-up at week1, month3, month6
  Number of Participants with diagnosed through a physical examination showing a hard lump, bruising, abnormal skin color, and subcutaneous hemorrhage, sometimes with shallow rugae in the scrotum
Hernia recurrence | post-operative follow-up at month3, month6
  Number of Participants with diagnosed through a physical examination showing intermittent bulge in the groin and can not get above mass
Testicular atrophy | post-operative follow-up at month3, month6
  Number of Participants with the testicular volume is reduced by 20% from pre- to post-operation after measuring the width, length and height of the testicles in centimeters, it is considered testicular atrophy.

SECONDARY OUTCOMES:
Course of pain killer requirement | post-operative follow-up at week1
  Measures the amount of painkiller medication used for less than or equal to 1 day or more than 1 day.

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi hospital, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cirocchi R, Popivanov GI, Cianci MC, Morabito A, Matteucci M, Lauricella S, Cassini D, Boselli C, Szergyuk I, Tebala GD, Rizzuto A, Bruzzone P. Comparison of Hernia Sac Transection and Full Sac Reduction for the Treatment of Inguinal Hernias: A Systematic Review and Meta-Analysis of Clinical Trials. World J Surg. 2025 Mar;49(3):590-604. doi: 10.1002/wjs.12474. Epub 2025 Jan 24. PMID 39856021
- [Result] Al-Taher RN, Khrais IA, Alma'aitah S, Al Saiad AA, Al-Abboodi AA, Saleh OM, Dwekat N, Almaaitah HW, Bello ZM, Rashdan MZ. Is the open approach superior to the laparoscopic hernia repair in children? A retrospective comparative study. Ann Med Surg (Lond). 2021 Sep 22;71:102889. doi: 10.1016/j.amsu.2021.102889. eCollection 2021 Nov. PMID 34691442
- [Result] Esposito C, Escolino M, Turra F, Roberti A, Cerulo M, Farina A, Caiazzo S, Cortese G, Servillo G, Settimi A. Current concepts in the management of inguinal hernia and hydrocele in pediatric patients in laparoscopic era. Semin Pediatr Surg. 2016 Aug;25(4):232-40. doi: 10.1053/j.sempedsurg.2016.05.006. Epub 2016 May 11. PMID 27521714
- [Result] Kevin E, Chukwubuike K. Complications of inguinal hernia repair in children: A tertiary hospital experience. Journal of Kathmandu Medical College. 2021;9.
- [Result] Aihole JS. The demographic profile and the management of infantile inguinal hernia: a 3-year's review. African Journal of Urology. 2020;26(1):28.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT07252999/Prot_SAP_000.pdf